CLINICAL TRIAL: NCT00919321
Title: The Duration of Humoral Immunity and the Memory Cell Function After Vaccination With 7-valent Pneumococcal Conjugate Vaccine in CLL
Acronym: KLL2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, MSinisalo, Dr, Tampere University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R09082M; 2009-012099-29 (EudraCT Number)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: CLL; PPV; PCV
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PPV (Other)
  Interventions: Biological: Pneumococcal polysaccharide vaccine (PPV)

INTERVENTIONS:
Biological: Pneumococcal polysaccharide vaccine (PPV) — One intramuscular injection

SUMMARY:
Patients with chronic lymphocytic leukemia (CLL)have had very poor humoral responses to pneumococcal polysaccharide vaccine (PPV). The vaccine in which pneumococcal polysaccharide antigens are conjugated to protein (PCV) have been immunogenic in CLL patients in our previous studies.

The purpose of this study is to evaluate the duration of these vaccine-induced antibodies and the function of memory cells by giving a one dose of PPV-vaccine after several years of PCV-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* CLL patients and controls who have been vaccinated with PCV in our previous study

Exclusion Criteria:

* Vaccinated with PPV-vaccine within the last 5 years, immunoglobulin substitution, corticosteroid treatment (equivalent of 20mg prednisolone per day)

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Antibody response | 1-3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Background] Sinisalo M, Vilpo J, Itala M, Vakevainen M, Taurio J, Aittoniemi J. Antibody response to 7-valent conjugated pneumococcal vaccine in patients with chronic lymphocytic leukaemia. Vaccine. 2007 Dec 21;26(1):82-7. doi: 10.1016/j.vaccine.2007.10.053. Epub 2007 Nov 12. PMID 18053620
- [Background] Sinisalo M, Aittoniemi J, Oivanen P, Kayhty H, Olander RM, Vilpo J. Response to vaccination against different types of antigens in patients with chronic lymphocytic leukaemia. Br J Haematol. 2001 Jul;114(1):107-10. doi: 10.1046/j.1365-2141.2001.02882.x. PMID 11472353
- [Derived] Lindstrom V, Aittoniemi J, Salmenniemi U, Kayhty H, Huhtala H, Itala-Remes M, Sinisalo M. Antibody persistence after pneumococcal conjugate vaccination in patients with chronic lymphocytic leukemia. Hum Vaccin Immunother. 2018 Jun 3;14(6):1471-1474. doi: 10.1080/21645515.2018.1436424. Epub 2018 Feb 23. PMID 29420116